CLINICAL TRIAL: NCT00775489
Title: The Effect of Beclomethasone Nasal Spray on Intraocular Pressure in Ocular Hypertension or Controlled Glaucoma
Brief Title: Nasal Steroids in Controlled Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Glaucoma Research Society of Canada (Other)
Responsible Party: Graham Trope / Professor, University of Toronto
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UHNToronto001
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2008-10

CONDITIONS: Intraocular Pressure
Keywords: glaucoma, steroid, nasal
MeSH Terms: conditions — Glaucoma | interventions — Beclomethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Steroid nasal spray (beclomethasone)
  Interventions: Drug: Nasal steroid Beclomethasone
- 2 (Placebo Comparator): Normal saline nasal spray
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Nasal steroid Beclomethasone — Beclomethasone nasal steroids to be given to a very well controlled glaucoma patients to find if this normal dose will lead to increase in intraocular pressure up to 20% where the study will be stopped at this point.
  Other Names: Beconase
  Arms: 1
Drug: Saline — control group will receive normal saline inhaler
  Arms: 2

SUMMARY:
Patients that have consented to participate in the study will be randomly assigned to one of two groups: control group or nasal steroid group. Patients in the control group will receive normal saline inhaler. Patients in the study group will receive steroid inhaler Follow-up visits are: baseline and weeks 2, 4, 6 after starting the spray. Intraocular pressure will be recorded on all visits.

DETAILED DESCRIPTION:
Systemic and topical ophthalmic steroids have long been associated with ocular effects, such as glaucoma or cataracts. Periocular steroid injections and steroids applied to periocular skin have also been reported to increase intraocular pressure (IOP) and raised IOP is the major risk factor for glaucoma. Approximately 18 to 36% of the general population are corticosteroid responders. This response is increased to 46 to 92% in patients with primary open-angle glaucoma (POAG).

Allergic rhinitis affects up to 30% of adults and 40% of children in the United States. Topical nasal steroids are the most effective treatment option.Nonallergic rhinitis is a common disease that affects approximately 17 million persons in the United States; approximately 22 million have a combination of allergic and nonallergic rhinitis.Topical nasal steroids have demonstrated efficacy in the treatment of nonallergic rhinitis and are considered first-line empiric therapy.With the perceived safety of nasal steroids, their use for the treatment of upper respiratory allergy has become more common.However, inhaled and nasal steroids might be absorbed systemically. Although the systemic absorption of inhaled and nasal steroids has been established, the clinically relevant ocular side effects are poorly defined. A large prospective study in 1995 by Samiy et al reported no statistically significant increase of IOP in 187 patients without glaucoma taking inhaled steroids for various pulmonary conditions. Similarly, a large case-control study in 1997 cases suggested that the presence of nasal steroid use in patients with newly diagnosed glaucoma or OHT versus nonglaucomatous patients was not statistically significant (odds ratio, 1.02; 95% CI, 0.59-1.77). However, the number of patients taking continuous high-dose nasal steroids was too small for statistical analysis. In 1998, a small prospective study of 26 non-glaucomatous patients revealed no evidence of OHT or cataracts after prolonged use of nasal steroids after endoscopic sinus surgery (mean follow-up, 8.8 ± 3.6 months; range, 3-19 months). A study of 61 patients with seasonal allergic rhinitis taking nasal fluticasone for 1 year showed no increased risk for glaucoma.However, no information was described regarding their glaucoma risk status before steroid use in this study. Six cases of increased IOP associated with combined nasal and inhaled steroid use in non-glaucomatous patients have been reported.

Considering the large number of patients on nasal steroids; It is surprising that no one has investigated if nasal steroid use is contraindicated in glaucoma patients.

ELIGIBILITY:
Inclusion criteria included the following:

* age 18 to 85 years inclusive
* OHT or mild to moderate POAG with cup-disc ratio of less than 0.8 vertically and mean deviation of less than -12.00 dB on Humphrey perimetry
* well controlled disease defined by IOP being at target and no visual field or disc progression for a minimum of 6 months

Exclusion criteria included the following:

* any form of steroid medication use within the last 6 weeks
* previous intra-ocular or refractive surgery
* no light perception vision.

Patients with or without rhinitis (allergic/ non-allergic/ mixed), with rhinitis defined as allergies and/ or nasal congestion present for greater than one year, were eligible.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Statistical analysis of associations between nasal corticosteroid use and elevated IOP | : 6 weeks from the beginning of treatment or IOP change by ≥ 20%.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Trope, Professor, Principal Investigator — University Health Network, Toronto
Locations (1):
- University of Toronto; Toronto Western Hospital, Toronto, Ontario, Canada